CLINICAL TRIAL: NCT03174405
Title: Avelumab and Cetuximab in Combination With FOLFOX in Patients With Previously Untreated Metastatic Colorectal Cancer - The Phase II AVETUX- Colorectal Cancer (CRC) Trial.
Brief Title: Avelumab and Cetuximab in Combination With FOLFOX in Patients With Previously Untreated Metastatic Colorectal Cancer - The Phase II AVETUX-CRC Trial.
Acronym: AVETUX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KRK-0216; 2016-004434-26 (EudraCT Number); MS100070_0065 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AVELUMAB (Experimental)
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — All eligible patients will receive cetuximab and mFOLFOX6 combined avelumab from the second cycle onwards.
  Cetuximab at a dose of 250 mg/m2 IV over 60 to 90 min (day 1 and 8) (first dose 400mg/m2) mFOLFOX6 (administration according to local standard) Oxaliplatin at a dose of 85 mg/m2 IV (day 1) 5-FU 400 mg/m2 IV bolus (day 1) LV at a dose of 400 mg/m2 iv (day 1) 5-FU at a dose of 2400 mg/m2 IV (day 1-3) Avelumab at a dose of 10mg/kg IV over 60 to 90 min (day 1 from cycle 2 onwards)

SUMMARY:
AVETUX is a single arm multicentric phase II investigator initiated trial conducted by the Arbeitsgemeinschaft Internistische Onkologie (AIO) in 11 German sites in patients with previously untreated RAS/BRAF wildtype mCRC independent of MSI status.

DETAILED DESCRIPTION:
The primary clinical objective is to determine the efficacy of a standard 1st line regimen (FOLFOX and cetuximab) in patients with RAS/v-Raf murine sarcoma viral oncogene homolog B (BRAF) wildtype, Microsatellite Instability (MSI) or icrosatellite Stability (MSS) MCRC with avelumab in terms of progression free survival rate after 12 months (acc. to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1).

The main secondary objective is to determine safety and tolerability, according to NCI Common Terminology Criteria for Adverse Events (CTCAE v4.03) and to the obtained data on vital signs, clinical parameters (oxygen saturation) and feasibility of the regimen. Further secondary objectives are to determine the efficacy of the experimental regimen in terms of objective response rate (acc. to RECIST v1.1 and irRECIST), and overall survival, to correlate clonal dynamics (RAS/EGFR subclones) with immune response signature to determine control of mutant subclones by the combination of anti-Epidermal growth factor receptor (EGFR) with anti-PD-L1and PD-L1 staining (and MSI status) with efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed, previously untreated RAS and BRAF wildtype, MSI or MSS metastatic colorectal cancer (primary tumor may be present)
2. Patients with at least one measurable lesion acc. to RECIST v1.1
3. ECOG Performance status ≤ 1
4. Life expectancy > 3 months
5. Age ≥ 18 years.
6. Haematologic function as follows: ANC ≥ 1.5 x 10^9/L, platelets ≥ 100 x10^9/L, hemoglobin ≥ 9 g/dL or 5.59 mmol/L
7. Adequate liver function as measured by serum transaminases (AST & ALT) ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN) and total bilirubin ≤ 1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled.
8. Adequate renal function: serum creatinine ≤ 1.5 x ULN
9. Negative serum pregnancy test at screening for women of childbearing potential. 10. Highly effective contraception for both male and female subjects if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1 % per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 90 days after avelumab treatment and 6 month after standard chemotherapy.

11. At least 6 months after completion of adjuvant chemotherapy. 12. Written informed consent 13. Ability to comply with the protocol for the duration of the study, including hospital/office visits for treatment and scheduled follow-up visits and examinations

Exclusion Criteria:

1. Malignancies other than disease under study within 5 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
2. All subjects with known brain metastases, except those meeting the following criteria:

   1. Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrolment
   2. No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
   3. Subjects must be either off steroids or on a stable or decreasing dose of <10mg daily prednisone (or equivalent)
3. Prior organ transplantation, including allogeneic stem-cell transplantation
4. Significant acute or chronic infections including, among others:

   1. Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
   2. Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
5. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent (Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible)
6. Concomitant treatment with corticosteroids or other immunosuppressants, besides treatment of brain metastases as mentioned in criteria 2 or:

   1. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
   2. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
7. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
8. Pregnancy or lactation
9. Known alcohol or drug abuse 10. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.

11. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.

12. All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma, colitis and pneumonitis), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment 13. Any psychiatric condition that would prohibit the understanding or rendering of informed consent 14. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines 15. Any approved anticancer therapy, including chemotherapy, hormonal therapy or radiotherapy, within 4 weeks prior to initiation of study treatment 16. Major surgical procedure within 28 days prior to treatment or anticipation of need for a major surgical procedure during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival Rate (PFS) @ 12 months | during 12 months of treatment
  PFS according to RECIST 1.1 at 12months of treatment

SECONDARY OUTCOMES:
Safety | 21 months
  Safety and tolerability (acc. to NCI CTC AE v4.03 and to the obtained data on vital signs, clinical parameters (oxygen saturation) and feasibility of the regimen)
Response Rate (RR) | 4 years
  Response Rate (RR) according to RECIST v1.1 and modified RECIST (mRECIST)
Progression Free Survival (PFS) | 4 years
  Progression Free Survival (PFS) according to RECIST v1.1 and mRECIST
Overall survival (OS) | 4 years
  Overall survival (OS)
Translational research | 48 months
  Translational research (correlation of clonal dynamics (RAS/EGFR subclones) with immune response signature to determine control of mutant subclones by the combination of anti-EGFR with anti-PD-L1, and PD-L1 (and MSI) status with efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stein, PD Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tintelnot J, Ristow I, Sauer M, Simnica D, Schultheiss C, Scholz R, Goekkurt E, von Wenserski L, Willscher E, Paschold L, Lorenzen S, Riera-Knorrenschild J, Depenbusch R, Ettrich TJ, Dorfel S, Al-Batran SE, Karthaus M, Pelzer U, Hinke A, Bauer M, Massa C, Seliger B, Wickenhauser C, Bokemeyer C, Hegewisch-Becker S, Binder M, Stein A. Translational analysis and final efficacy of the AVETUX trial - Avelumab, cetuximab and FOLFOX in metastatic colorectal cancer. Front Oncol. 2022 Dec 20;12:993611. doi: 10.3389/fonc.2022.993611. eCollection 2022. PMID 36605436
- [Derived] Stein A, Simnica D, Schultheiss C, Scholz R, Tintelnot J, Gokkurt E, von Wenserski L, Willscher E, Paschold L, Sauer M, Lorenzen S, Riera-Knorrenschild J, Depenbusch R, Ettrich TJ, Dorfel S, Al-Batran SE, Karthaus M, Pelzer U, Waberer L, Hinke A, Bauer M, Massa C, Seliger B, Wickenhauser C, Bokemeyer C, Hegewisch-Becker S, Binder M. PD-L1 targeting and subclonal immune escape mediated by PD-L1 mutations in metastatic colorectal cancer. J Immunother Cancer. 2021 Jul;9(7):e002844. doi: 10.1136/jitc-2021-002844. PMID 34315821
- See also: Homepage of the AIO (Arbeitsgemeinschaft Internistische Onkologie in der Deutschen Krebsgesellschaft e.V.) — http://www.aio-portal.de/